CLINICAL TRIAL: NCT00496418
Title: Randomized Controlled Open Interventional Study for Evaluation of Use of Peristomal Mesh for Prophylaxis of Parastomal Hernia
Brief Title: Peristomal Mesh for Prophylaxis of Parastomal Hernia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Jan Lambrecht, MD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-07203a
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Hernia
Keywords: colostomy; parastomal; peristomal; hernia; mesh; surgery; Indication for permanent end colostomy
MeSH Terms: conditions — Hernia

ARMS (2):
- Prophylactic stoma mesh (Experimental): Mesh
  Interventions: Device: Mesh in permanent colostomy
- No mesh prophylaxis (Active Comparator): No mesh
  Interventions: Device: Mesh in permanent colostomy

INTERVENTIONS:
Device: Mesh in permanent colostomy

SUMMARY:
The study aims to prove differences or equalities in outcome for patients operated with or without a peristomal mesh in the sublay position when establishing a permanent colostomy.

DETAILED DESCRIPTION:
Patients are randomized to 2 groups equal in number: a group with mesh implantation and a control group without mesh implantation.

Primary endpoint is Parastomal hernia. Secondary endpoints are operating time, infection, obstruction, stenosis, retraction, fistulae, skin related problems and reoperations. Endpoints are correlated to body mass index, previous hernia, age, concurrent illness and cause for colostomy. Patients are followed 4 years after operation with clinical examination

ELIGIBILITY:
Inclusion Criteria:

* Condition with indication for establishing a permanent end-colostomy.

Exclusion Criteria:

* Age under 18
* ASA score above 3

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-07; Primary Completion 2011-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Parastomal hernia | at 3, 12, 24, 36 and 48 months

SECONDARY OUTCOMES:
Operating time, infection, obstruction, stenosis, retraction, fistulae, skin related problems and reoperations. Endpoints are correlated to body mass index, previous hernia, age, concurrent illness and cause for colostomy | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan Lambrecht, MD, Principal Investigator — Rikshospitalet-Radiumhospitalet HF, Medical Center
Locations (1):
- Rikshospitalet-Radiumhospitalet HF, Oslo, Norway

REFERENCES:
- [Derived] Lambrecht JR. Diagnostic methods in parastomal hernia; research and clinical relevance. Hernia. 2021 Jun;25(3):817-820. doi: 10.1007/s10029-020-02177-8. Epub 2020 Mar 28. No abstract available. PMID 32222841